CLINICAL TRIAL: NCT03232697
Title: French Language Validation of the Phone Version of the Montreal Cognitive Assessment (MoCA)
Brief Title: French Language Validation of the 5-minutes Montreal Cognitive Assessment (MoCA)
Acronym: MoCATEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016_47; 2017-A00131-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-07-21; First posted 2017-07-28 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-08

CONDITIONS: Cognitive Symptom; Evaluations, Diagnostic Self
MeSH Terms: conditions — Neurobehavioral Manifestations

STUDY DESIGN:
Intervention Model Description: Different populations including subjects with or without cognitive impairment will be used to determine the accuracy of a short version of the MOCA as compared to the full version of this scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy subjects (Other): Subjects will be submitted to both the full version of the Montreal Cognitive Assessment and of the 5-minutes version of the Montreal Cognitive Assessment
  Interventions: Diagnostic Test: Full version of the Montreal Cognitive Assessment; Diagnostic Test: 5 minutes version of the Montreal Cognitive Assessment
- Alzheimer patients (Other): Patients will be submitted to both the full version of the Montreal Cognitive Assessment and of the 5-minutes version of the Montreal Cognitive Assessment
  Interventions: Diagnostic Test: Full version of the Montreal Cognitive Assessment; Diagnostic Test: 5 minutes version of the Montreal Cognitive Assessment
- Parkinson and Huntington patients (Other): Patients will be submitted to both the full version of the Montreal Cognitive Assessment and of the 5-minutes version of the Montreal Cognitive Assessment
  Interventions: Diagnostic Test: Full version of the Montreal Cognitive Assessment; Diagnostic Test: 5 minutes version of the Montreal Cognitive Assessment
- Diabetic patients (Other): Patients will be submitted to both the full version of the Montreal Cognitive Assessment and of the 5-minutes version of the Montreal Cognitive Assessment
  Interventions: Diagnostic Test: Full version of the Montreal Cognitive Assessment; Diagnostic Test: 5 minutes version of the Montreal Cognitive Assessment

INTERVENTIONS:
Diagnostic Test: Full version of the Montreal Cognitive Assessment — Patients or subjects will be submitted to the full version of the MOCA
Diagnostic Test: 5 minutes version of the Montreal Cognitive Assessment — The same patients and subjects will be submitted to the 5 minutes version of the MOCA through a phone call

SUMMARY:
The aim of the study is to validate a french version of the 5 minutes version of the Montreal Cognitive Assessment as compared to the french full version of this test.

DETAILED DESCRIPTION:
The Montreal Cognitive Assessment (MOCA) is a test used to detect cognitive impairments. This test is available in different languages including french. A short version (the 5 minutes MOCA) has also been validated through a phone call use that allows to develop some epidemiological approaches. Nevertheless, this short version has not been validated in french.

The main aim of the study is to validate the french translation of the short version of the MOCA as compared the the full french version of the test.

To validate the short version, several groups of subjects will be included : healthy subjects, Alzheimer disease patients, Parkinson or Huntington diseases patients as well as diabetic patients.

The inclusion of both healthy subjects and patients with different types of cognitive impairments will allow to validate the short version of the test.

All subjects and patients will first be submitted to the full version of the MOCA during a face to face procedure. Thirty to forty days later, they will be submitted to the short version of the test through a phone call performed by an independent rater.

Subgroups of healthy subjects and patients will also be used to determine the test-retest and inter-rater reliability of the short version of the MOCA.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers

* Volunteers, BMI <26
* free from neurological, psychiatric, metabolic or cardiac pathologies;
* Absence of active metabolic or cardiac diseases, unstabilized under treatment
* Pregnant test negative

Patients

* Patients suffering from pathologies that may be accompanied by cognitive decline or dementia (Alzheimer's disease, Parkinson's and Huntington's disease, diabetes) that meet the usual diagnostic criteria for these diseases;
* Patients should not start treatment of a new therapeutic class under test

Exclusion Criteria:

* Pregnant or nursing women.
* Illiterate subjects
* Presence of uncorrected visual or auditory disturbances
* "Alcohol use disorder" observed at the Mini International Neuropsychiatric Inventory (MINI);
* "Substance use disorder" observed at the MINI;
* Participation in a therapeutic trial or in an exclusion period from a previous clinical trial;
* Patient whose physical or mental condition does not allow them to pass the study tests;
* Persons under guardianship or under trusteeship;
* Recent cognitive assessment (less than 6 months) by the classic MoCA

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Correlation between scores obtained with the different versions of the MOCA | 30 to 40 days
  To measure the correlation between the results obtained at the short and full versions of the MOCA

SECONDARY OUTCOMES:
Performance of the short version of the MOCA | 30 to 40 days
  Receiver operator characteristic (ROC) analyses of the short version of MOCA to determine cognitive impairment as compared to full version as a gold-standard
Test-retest reliability | 30 to 40 days
  To determine the test-retest reliability of the short version of the MOCA
Inter-rater reliability | 30 to 40 days
  To determine the inter-rater reliability of the short version of the MOCA

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Deplanque, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- University Hospital, Lille, France

IPD SHARING:
Plan to Share IPD: No